CLINICAL TRIAL: NCT03388814
Title: Speeding Recovery From Pain and Opioid Use After Mastectomy and Breast Reconstruction Surgery
Brief Title: Speeding Recovery From Pain and Opioid Use
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00047335
Record Dates: First submitted 2017-12-19; First posted 2018-01-03 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Pain, Postoperative; Breast Cancer; Opioid Use; Surgery
Keywords: PPBCS; Acute; Postoperative; Mastectomy; Breast Reconstruction
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine Group (Active Comparator): Those patients randomized to surgeon infiltration will have a skin wheal performed with lidocaine at the site where an actual pectoralis nerve block would be performed as visualized using ultrasound. Surgeons performing infiltration techniques will be blinded to the contents of the injectate and those patients randomized to surgeon infiltration will receive pharmacy study drug labeled bupivacaine injected in the same fashion and volume as the saline group for oncologic and plastic surgery.
  Interventions: Drug: Local infiltration of bupivacaine
- Pectoralis Nerve block Group (Experimental): Those patients who are randomized to pectoralis nerve block will have randomization immediately preoperatively and will undergo the nerve block procedure using local anesthetic in the standard fashion. Those patients randomized to pectoralis block will have a standard volume of normal saline injected for oncologic and plastic surgery.
  Interventions: Drug: Pectoralis Nerve block

INTERVENTIONS:
Drug: Local infiltration of bupivacaine — Patients assigned to the local infiltration with bupivacaine group will receive 30 ml of 0.25% bupivacaine with 1:200,000 epinephrine. These injections will occur at the end of the mastectomy and prior to the insertion of the tissue expander implant. The local anesthetic will be injected into the chest wall and skin flaps. Attending physicians and resident physicians will receive prior instruction regarding correct placement of the local anesthetic so that it will be consistently placed in the same locations with similar volume distribution.
  Arms: Bupivacaine Group
Drug: Pectoralis Nerve block — Patients assigned to the pectoralis block group will receive a total of 20 ml 0.25% bupivacaine (with 1:200,000 epinephrine and 1.67 mcg clonidine per ml) in the tissue plane between the serratus anterior and the pectoralis minor muscles at approximately the level of the 4th rib and 10 ml of the same solution in the tissue plane between the two pectoralis muscles at approximately the 3rd rib under ultrasound guidance on the surgical side preoperatively.
  Arms: Pectoralis Nerve block Group

SUMMARY:
Surgical treatment of breast cancer is associated with significant disability, and pain is often reported as a primary cause for declines in the ability to perform activities of daily living. However, breast reconstruction at the same time as mastectomy has been linked to higher postoperative pain, which can be a risk factor for persistent pain. The goal of this study is to determine the speed of recovery from pain and opioid use in the first 2 months after breast surgery and reconstruction.

DETAILED DESCRIPTION:
Surgical treatment of breast cancer is associated with significant disability, and pain is often reported as a primary cause for declines in the ability to perform activities of daily living. Surgical treatments can also negatively influence social exposure and alter self-perception and sexual health. Reconstruction of the breast mound following mastectomy has several benefits in psychosocial functioning, body image and satisfaction with breast appearance, and sexual well-being. However, reconstruction at the same time as mastectomy has been linked to higher postoperative pain. Compared to autologous breast reconstruction, implant based techniques have been linked to higher requirements of postoperative nonsteroidal anti-inflammatory drugs, opioids, and benzodiazepines as well as higher pain scores in the immediate postoperative period and one year after surgery. Recent publications report that intensity of pain in the operative area prior to surgery, body mass index (BMI), presence of axillary operation, intensity of acute postoperative pain, and amount of opioid required to achieve satisfactory analgesia in the acute postoperative period are also risk factors for persistent pain following breast cancer surgery (PPBCS). Since severity of acute postoperative pain is consistently observed as a risk factor for persistent pain, there has been interest in determining whether better acute pain control reduces this risk. Infiltration of the surgical site with bupivacaine decreases intraoperative and postoperative narcotic use, and has been associated with decreased pain scores in the immediate postoperative period. A novel approach to hemithoracic analgesia has been introduced which proposed less risk of anatomic trespass by doing a local anesthetic injection into the fascial planes of the chest wall. These procedures have demonstrated improved analgesia for breast surgeries. Unfortunately, there is a lack of large, multicenter, prospective, and randomized trials comparing these analgesic modalities and evaluating the response to these acute postoperative analgesic interventions with regard to PPBCS and other metrics of daily function, satisfaction with pain control, and self-perception of well-being and predictors of recovery from the pain state. The goals of this research are to provide short-term surrogate measures for prevention or treatment trials and to develop methods enabling practitioners to forecast recovery in real-time and that are translatable to patients in understandable references regarding risk over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unilateral mastectomy with immediate issue expander and implant based reconstruction.
* Age ≥ 18 years
* Ability to understand, read, and write English, and the willingness to sign an IRB-approved informed consent document.
* Patients who receive a tissue expander placement will be included in the study.
* American Society of Anesthesiologists physical status I-III patients.

Exclusion Criteria:

* Patients who receive an autologous tissue reconstruction.
* Patients who receive a bilateral reconstruction.
* Patients who receive a direct to permanent implant reconstruction
* Patients with diagnosis of opioid misuse disorder or on high dose opioid therapy (greater than 100 mg equivalents of oral morphine per day)
* Patients who are wards of the state
* Patients who cannot read or speak English
* History of allergic reactions attributed to compounds with known or suspected cross-sensitivity to bupivacaine.
* Pregnant or breast feeding
* Inability to access to the internet on a daily basis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Modeled worst pain intensity using the numeric rating scale (NRS) | From study start to 2 months after surgery
  NRS pain scores will be obtained daily from time of initiation into the study until 2 months after surgery and the scores following hospital discharge will be modeled for each individual using a growth curve change-point approach. The NRS has a 0-10 numeric rating scale (0=no pain and 10=worst pain imaginable), where lower scores denotes better outcomes.

SECONDARY OUTCOMES:
Area under the curve of the numeric rating scale (NRS) | During the first 48 hours postoperatively
  The NRS has a 0-10 numeric rating scale (0=no pain and 10=worst pain imaginable), where lower scores denotes better outcomes.
Opioid use | From admission to 2 months after surgery
  Opioid use converted to morphine equivalents while in hospital and daily for the first 2 months after surgery
Length of stay for hospitalization | At Discharge (up to 30 days)
  Length of stay for hospitalization after mastectomy and breast reconstruction. Time is counted from admission to hospital discharged.
Readmission rates | 6 months after mastectomy and breast reconstruction
  Readmission rates to the hospital within 6 months after mastectomy and breast reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Doug Jaffe, DO, Principal Investigator — Wake Forest University Health Sciences